CLINICAL TRIAL: NCT01068249
Title: A Phase II Study of Letrozole and RAD001 (Everolimus) in Patients With Advanced or Recurrent Endometrial Cancer
Brief Title: Letrozole and RAD001 With Advanced or Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0059; NCI-2011-03639 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer
Keywords: Advanced; Recurrent; Progressive; Endometrial Cancer; Letrozole; RAD001; Afinitor; Everolimus; Femara
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — Letrozole; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letrozole + RAD001 (Experimental): Letrozole and RAD001 (Everolimus)
  Interventions: Drug: Letrozole; Drug: RAD001 (Everolimus)

INTERVENTIONS:
Drug: Letrozole — 2.5 mg daily by mouth every day, at same time as Everolimus.
  Other Names: Femara
Drug: RAD001 (Everolimus) — 10 mg by mouth daily
  Other Names: Afinitor

SUMMARY:
The goal of this clinical research study is to learn if the combination of RAD001 (everolimus) and Femara (letrozole) can help to control recurrent or progressive endometrial cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Everolimus is designed to stop cancer cells from multiplying. It may also stop the growth of new blood vessels that help tumor growth, which may cause the tumor cells to die.

Letrozole is designed to block chemical pathways that are necessary for tumor growth.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 2 pills of everolimus by mouth 1 time every day. You should not open everolimus until you are about to take it because it absorbs moisture and is sensitive to light. You will also take 1 pill of letrozole by mouth 1 time every day. You should take letrozole at the same time as everolimus.

Everolimus should be taken the same time every day on an empty stomach (fasting state) or after no more than a light, fat-free meal. You should wait at least 6 hours after a eating a regular (not fat-free meal) before taking everolimus. You should not eat fatty foods for at least 1 hour after taking everolimus.

If you cannot swallow the tablets, the tablets should be dissolved in a glass of about 2 tablespoons of water just before being taken. The tablets should then be stirred gently (for a maximum of 7 minutes) until the tablets are dissolved. The contents should then be drunk. If you vomit after taking the study drug, you should not take another tablet that day. If you forgot to take the drug one day, you should not take an extra dose the next day but instead contact your doctor for advice.

You will be given a diary where you will record the pills you take each day. You must bring this diary to each visit.

While you are on study, you should avoid grapefruit, grapefruit juice, and other products containing grapefruit. There are also certain drugs you cannot take during this study. You should not take any drugs during the study without asking the study doctor first.

Study Visits:

Every 4 weeks, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs (blood pressure, heart rate, breathing rate, and temperature).
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests, including checking your liver and kidneys and measuring the levels of sugar in your blood, and levels of fat in your blood.
* You will asked about any side effects you have experienced.
* If the disease is in the pelvis, you will have a pelvic exam.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn for hepatitis testing.
* Your pills will be counted.

At Week 8, the following tests and procedures will be performed:

* You will have a physical exam, including a pelvic exam.
* You will have a CT and/or MRI scan of your chest, abdomen, and pelvis. Other areas will be scanned if the doctor thinks it is needed.
* Any tumors will be measured. The doctor will either feel the tumor or a CT, x-ray, and/or MRI will be used.
* If the disease is in your chest, you will have chest CT and/or MRI scan to check the status of the disease.
* You will asked about any side effects you have experienced.

After the Week 8 Visit, you will have the following tests and procedures. (If the disease has partially or completely responded to the study drugs, these tests will be done around Week 12. If the disease is stable, these tests will be done around Week 16.)

* You will have a physical exam.
* You will have a CT and/or MRI scan of your chest, abdomen, and pelvis. Other areas will be scanned if the doctor thinks it is needed.
* Any tumors will be measured. The doctor will either feel the tumor or a CT scan, x-ray, and/or MRI will be used.
* If the disease is in your chest, you will have a chest CT and/or MRI scan to check the status of the disease.

After the Week 12 or 16 visit, every 12 weeks, the following tests and procedures will be performed:

* You will have a pelvic exam.
* You will have a CT and/or MRI scan of your chest, abdomen, and pelvis. Other areas will be scanned if the doctor thinks it is needed.

I-f the disease is in your chest, you will have chest CT and/or MRI scan to check the status of the disease.

Length of Study:

You may continue receiving additional cycles of study treatment. You will be taken off study if you experience intolerable side effects, the disease gets worse, the disease completely responds, or the doctor thinks it is in your best interest.

End of Treatment Visit:

Within 4 weeks after the last dose of study drugs, you will have an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a pelvic exam.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests, including checking your liver and kidneys and measuring the levels of sugar in your blood, and levels of fat in your blood.
* You will have a CT and/or MRI scan of your chest, abdomen, and pelvis. Other areas will be scanned if the doctor thinks it is needed.
* If the disease is in your chest, you will have chest CT and/or MRI scan to check the status of the disease.
* Your pills will be counted and any unused study drug will be returned.

Long Term Follow-up:

After you are off study, you will be followed by your doctor on a regular basis. How often these visits occur are up to you and your doctor. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will have a pelvic exam.
* Your performance status will be recorded.
* You will be asked if you have experienced any intolerable side effects.
* You will have a CT and/or MRI scan of your chest, abdomen, and pelvis. Other areas will be scanned if the doctor thinks it is needed.
* If the disease is in your chest, you will have chest CT and/or MRI scan to check the status of the disease.

This is an investigational study. Everolimus is not FDA approved or commercially available. At this time, everolimus is only being used in research. Letrozole is FDA approved and commercially available for the treatment of breast cancer and ovarian cancer. The combination of everolimus and letrozole in this study for the treatment of endometrial cancer is also investigational. Up to 42 patients will take part in the multicenter study. Up to 42 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an approved informed consent.
2. Histologically confirmed endometrial cancer (endometrioid, serous, or clear cell, or mixed histology; any grade) which is considered progressive or recurrent.
3. Patients may have failed no more than two prior chemotherapeutic regimens for recurrent or advanced disease (including adjuvant therapy). Chemotherapy administered in conjunction with radiation as a radio-sensitizer is not counted as a prior treatment for recurrent or advanced disease.
4. All patients must have measurable disease as defined by RECIST 1.1.
5. Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST. Tumors within a previously irradiated field will be designated as "non-target" lesions, unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
6. Patients must have a Zubrod performance status of 0, 1, or 2.
7. Patients must not be of child bearing potential. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal for greater than 12 months. Patients in whom ovaries are present and were not previously menopausal at the time of hysterectomy, should have a serum estradiol < 10 pg/mL to confirm ovarian senescence.
8. Patients must have a pretreatment granulocyte count (i.e., segmented neutrophils + bands) of >1,500/Fl, a hemoglobin level of >/=9gm/dL and a platelet count of >100,000/Fl. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
9. Patients must have an adequate renal function of >50cc/min as documented by the Cockcroft Gault creatinine clearance formula: Estimated GFR = (140 - age) x (weight kg) divided by 72 x serum Creatinine (non-IDMS) x 0.85 (female)
10. Patients must have adequate hepatic function as documented by a serum bilirubin </=2.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor. Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
11. Alanine aminotransferase (SGPT) must be </= 3x institutional upper limit of normal unless the liver is involved with tumor, in that case, the alanine aminotransferase must be </= 5 x institutional upper limit of normal.
12. Prior to beginning therapy, at least 4 weeks must have elapsed since prior chemotherapy, surgery, radiation therapy, hormonal therapy or investigational therapy. Patients receiving palliative radiation therapy are exempt from the 4 week waiting period.
13. Baseline lipid levels (triglycerides, cholesterol) must be </= grade 1. Patients are allowed to be on lipid lowering drugs.
14. Patients must be >/= 18 years of age.

Exclusion Criteria:

1. Patients with intact ovarian function.
2. Patients who have previously received RAD001 or another mTOR inhibitor or letrozole or another aromatase inhibitor. Use of progestational or other hormonal agents are permitted provided they have not been administered within the previous 4 weeks.
3. Patients who have uterine sarcomas or mixed malignant mullerian tumors.
4. Patients who have isolated recurrences (vaginal, pelvic, or paraaortic) that are amenable to potentially curative treatment with radiation therapy or surgery.
5. Patients with any other severe concurrent disease, which would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
6. Patients currently receiving chemotherapy or radiotherapy or those in whom anti-cancer treatment has occurred within the preceding 4 weeks.
7. Chronic treatment with systemic steroids or another immuno-suppressive agent.
8. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period.
9. Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years
10. Patients with active infection that requires systemic antibiotics.
11. Patients with a known history of cardiac disease; i.e., uncontrolled hypertension (systolic B/P >/= 140 mm Hg and/or diastolic B/P >/= 90 mm Hg) or unstable angina. Patients with a history of myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, or symptoms suspicious for congestive heart failure are not eligible unless a left ventricular ejection fraction in the past 6 months is documented to be 50% or greater. Patients who have had a LVEF (performed for any reason) of less than 50% in the past 6 months are ineligible.
12. Patients with a known history severely impaired lung function (patients who are oxygen dependent).
13. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
14. Patients who are pregnant or breast-feeding.
15. Presence of clinically apparent untreated central nervous system metastases.
16. Patients with carcinomatous meningitis.
17. Patients with deep venous or arterial thrombosis (including pulmonary embolism) within 6 weeks of study entry. Patients may be on maintenance anticoagulation therapy.
18. Patients with previously documented human immunodeficiency virus (HIV) infection.
19. Patients with an impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-04-30 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2028-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela T. Soliman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Morristown Memorial Hospital, Women's Cancer Center, Morristown, New Jersey
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Slomovitz BM, Jiang Y, Yates MS, Soliman PT, Johnston T, Nowakowski M, Levenback C, Zhang Q, Ring K, Munsell MF, Gershenson DM, Lu KH, Coleman RL. Phase II study of everolimus and letrozole in patients with recurrent endometrial carcinoma. J Clin Oncol. 2015 Mar 10;33(8):930-6. doi: 10.1200/JCO.2014.58.3401. Epub 2015 Jan 26. PMID 25624430
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitments were done in a medical clinic setting.
Pre-assignment Details: 42 participants signed the consent, 3 participants were screen failures
Groups:
- RAD001 + Letrozole: RAD001 10 mg oral tablet daily + Letrozole 2.5 oral tablet daily for 28 days
Period: Overall Study
Arm/Group | RAD001 + Letrozole
Started | 39
Completed | 35
Not Completed | 4
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: All participants were included in the analysis
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 15
Age, Continuous [Median (Full Range); unit: years] | 59.9 [24 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Rate
Description: Objective response or stable disease rate monitored as patients accrue and are evaluated following the example of Thall and Simon. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: at 8 weeks of treatment, then every 12 weeks, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 35
Participants
  Complete Response (CR) | 9
  Partial Response (PR) | 2

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 30% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: from study entry (1st treatment) to date of tumor progression, date of death, or, for patients alive without tumor progression, date of last follow-up, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 35
months | 3 [1.9 to 15.7]

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact
Time Frame: from (1st treatment) to death or, for living patients, date of last contact, up to 24.4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 35
months | 14 [9.5 to 24.4]

4. Secondary Outcome: Number of Participants With Disease Progression
Time Frame: from study entry (1st treatment) to date of tumor progression, date of death, or, for patients alive without tumor progression, date of last follow-up, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 35
Participants | 31

5. Secondary Outcome: Number of Participants With Adverse Events (All Grades)
Description: Toxicity was assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 3.0).
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Letrozole
Number analyzed (Participants) | 35
Participants | 28

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment at 28 days plus 30 days post treatment, assessed up to 24.4 months
Arm/Group | RAD001 + Letrozole
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 28/35
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 + Letrozole (N=35)
Fatigue (General disorders) | 28
Hypertriglyceridemia (Metabolism and nutrition disorders) | 28
Hypercholesterolemia (Metabolism and nutrition disorders) | 27
Mucositis (Gastrointestinal disorders) | 25
Anemia (Blood and lymphatic system disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 21
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 10
Anorexia (Gastrointestinal disorders) | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Elevated AST (Investigations) | 2
Elevated ALT (Investigations) | 14
Hypomagnesemia (Investigations) | 13
Hypokalemia (Investigations) | 11
Diarrhea (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Edema: limbs (Blood and lymphatic system disorders) | 11
Headache (Nervous system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 13
Neuropathy- sensory (Nervous system disorders) | 12
Rash: acneiform (Skin and subcutaneous tissue disorders) | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Pruritus (Skin and subcutaneous tissue disorders) | 9
Taste alteration (Gastrointestinal disorders) | 9
Weight loss (Metabolism and nutrition disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 5
Chills (General disorders) | 5
Dizziness (Nervous system disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 6
Fever (General disorders) | 5
Hemorrhage - nasal (Respiratory, thoracic and mediastinal disorders) | 5
Insomnia (General disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nail Disorder (Skin and subcutaneous tissue disorders) | 6
Neutrophils decreased (Blood and lymphatic system disorders) | 5
Pain - extremities (Musculoskeletal and connective tissue disorders) | 7
Pain - other (Musculoskeletal and connective tissue disorders) | 5
Sweating (General disorders) | 7
Urinary Tract infection (Infections and infestations) | 5
Dry mouth (Gastrointestinal disorders) | 5
Alkaline phosphatase increased (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Auditory/ear (other) (Ear and labyrinth disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bladder pain (Hepatobiliary disorders) | 1
Blood/bone marrow (other) (Blood and lymphatic system disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Cardiac arrhythmia (other) (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dermatology/skin (other) (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Endocrine (other) (Endocrine disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
GI (other) (Gastrointestinal disorders) | 1
Infection (Infections and infestations) | 1
Infection (other) (Infections and infestations) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal sinus infection (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Serum glucose decreased (Metabolism and nutrition disorders) | 1
Serum potassium increased (Metabolism and nutrition disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Stomal ulcer (Injury, poisoning and procedural complications) | 1
Watering eyes (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT01068249/Prot_SAP_000.pdf